CLINICAL TRIAL: NCT06066580
Title: An Open-Label Extension Study to Assess the Long-term Effect of EDG-5506 on Safety, Biomarkers, and Functional Measures in Adults and Adolescents With Becker Muscular Dystrophy
Brief Title: Open-Label Extension of EDG-5506 in Participants With Becker Muscular Dystrophy
Acronym: MESA
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDG-5506-203
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Becker Muscular Dystrophy
Keywords: Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Drug: Sevasemten
  Interventions: Drug: Sevasemten

INTERVENTIONS:
Drug: Sevasemten — Sevasemten is administered orally once per day

SUMMARY:
EDG-5506-203 MESA is an open-label extension study to assess the long-term effect of sevasemten (EDG-5506) on safety, biomarkers, and functional measures in adults and adolescents with Becker muscular dystrophy

DETAILED DESCRIPTION:
This is an open-label, treatment extension study to evaluate the safety, tolerability, and durability of effect in long-term dosing of sevasemten. EDG-5506-203 MESA will provide continued access to sevasemten treatment to participants with Becker muscular dystrophy who were previously enrolled in EDG-5506-002 ARCH, completed EDG-5506-201 CANYON and GRAND CANYON, or completed EDG-5506-202 DUNE.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males with a diagnosis of BMD and participation in EDG-5506-002 ARCH, EDG-5506-201 CANYON and GRAND CANYON, or EDG-5506-202 DUNE. Participants are eligible if they complete the respective prior study visits as follows:

* EDG-5506-002 ARCH: Complete the final study Visit 27 [Month 24]; or, completion of the ET visit prior to Visit 27 [Month 24]
* EDG-5506-201 CANYON and GRAND CANYON: Complete the final study visit (Cohorts 1, 2, 4, and 5: Visit 12 [Month 12]; Cohort 6: Visit 11 [Month 18])
* EDG-5506-202 DUNE: Complete at least 36 weeks of open-label treatment (Visit 14 [Week 52])

Key Exclusion Criteria:

1. Any clinically significant changes during or following participation in EDG-5506-002, EDG-5506-201, or EDG-5506-202 that would affect the potential safety of the participant to receive sevasemten.
2. Receiving moderate or strong cytochrome P450 CYP3A4 inhibitors or inducers.
3. Receipt of an investigational drug other than sevasemten within 30 days or 5 half-lives (whichever is longer) of dosing in the present study.

3. Receipt of oral corticosteroids for the treatment of BMD in the previous 6 months.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events in those treated with sevasemten | 37 Months
Severity of adverse events in those treated with sevasemten | 37 Months

SECONDARY OUTCOMES:
Incidence of treatment-emergent abnormal clinical chemistry laboratory test results | 36 Months
Incidence of treatment-emergent abnormal hematology laboratory test results | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M. Donovan, MD, PhD, Study Chair — Edgewise Therapeutics, Inc.; Roxana D. Dreghici, MD, Study Chair — Edgewise Therapeutics, Inc.
Locations (46):
- United States (24):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC San Diego, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - UC Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Rare Disease Research, LLC NC, Hillsborough, North Carolina
  - University of Cincinnati Gardner Neuroscience Institute, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - National Neuromuscular Research Institute, Austin, Texas
  - Neurology Rare Disease Center, Denton, Texas
  - Virginia Commonwealth University Health, Richmond, Virginia
- Belgium (3):
  - University Hospital Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
  - Centre Hospitalier Régional de la Citadelle, Liége
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - Centre de Reference des Maladies Neuromusculaires et de la SLA - AP-HM Hopital de La Timone, Marseille
  - CHU de Nantes, Nantes
  - CHU de Nice - Hopital Pasteur 2 - Centre de reference des Maladies Neuromusculaires, Nice
  - AP-HP Hopital Pitie-Salpetriere, Paris
- Klinikum der Ludwig-Maximilians-Universitaet Muenchen, Munich, Germany
- Hadassah University Hospital, Jerusalem, Israel
- Italy (3):
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore, Milan
  - Azienda Ospedale - Università Padova, Padua
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - University College London Hospital, London
  - St. George's University Hospitals NHS Foundation Trust, London
  - Newcastle Freeman Hospital, Newcastle
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.edgewisetx.com